CLINICAL TRIAL: NCT00632060
Title: The Efficacy of Manual and Manipulative Therapy for Low Back Pain in Military Active Duty Personnel: A Feasibility Study
Brief Title: Manual and Manipulative Therapy for Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samueli Institute for Information Biology (Other)
Collaborators: Palmer Center for Chiropractic Research (PCCR) (Other); William Beaumont Army Medical Center (U.S. Federal Agency); United States Army Fort Bliss (Unknown)
Responsible Party: CPT Keith P. Myers, MC / Chief, WBAMC Physical Medicine and Rehabilitation, William Beaumont Army Medical Center (WBAMC)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1 EA-0000055; WBAMC #06/05; USUHS TX781-AX-2
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-02

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Manual / Manipulative Therapy
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

ARMS (2):
- 1 (No Intervention): Standard Care Control Group - Participants randomized to the standard care group will continue their use of non-prescription or prescription medication and reduced duty loads, as prescribed by the credentialed medical provider.
- 2 (Experimental): Manual / Manipulative Therapy Group: Participants randomized to the M/MT group will receive a course of M/MT along with standard care. The patient will see the chiropractor twice a week for the entire course of the study, regardless of manipulation or not.
  Interventions: Procedure: Manual / Manipulative Therapy (M/MT)

INTERVENTIONS:
Procedure: Manual / Manipulative Therapy (M/MT) — Subjects will receive M/MT twice a week for 4 weeks
  Other Names: M/MT
  Arms: 2

SUMMARY:
The specific aims of this research project are to determine feasibility of, and the comparative treatment effect size for, conducting a larger clinical trial of Manual/Manipulative Therapy (M/MT) in restoring peak performance in military personnel in operational environments and to evaluate the ability of the addition of M/MT to standard care to decrease pain and increase function for patients with low back pain.

The following two hypotheses will guide the data collection:

1. The primary hypothesis is that the addition of acourse of M/MT to standard care for low back pain will decrease pain at 4 weeks when compared to standard care alone
2. In addition, the secondary hypothesis will be that the addition of a course of M/MT to standard care for low back pain will decrease pain and increase function over 2 and 4 weeks when compared to standard care alone

DETAILED DESCRIPTION:
Musculoskeletal injuries are among the highest frequency injuries in military personnel(1). These may result from training exercises, normal job duties, or recreational activities (2). Such injuries may cause reduced levels of performance and therefore decrease military readiness (1). This prospective, randomized, clinical trial compares manual/manipulative therapy (M/MT) and standard care to standard care alone for episodes of low back pain. Patients will be randomized to standard care or standard care plus M/MT. Standard care consists of medication prescribed by the credentialed medical provider; M/MT will be delivered by the chiropractor physician. The trial time period will be 4 weeks with outcome measurements at intake, 2 weeks, and 4 weeks. Outcome measures include the Visual Analogue Scale (VAS) for pain, Roland-Morris Low Back Pain and Disability Questionnaire (RDQ), the Back Pain Functional Scale for assessing function (3), Global Improvement Questionnaire for patient perception regarding improvement in function, Patient Expectation and Patient Satisfaction Questionnaires to examine patient expectations toward care and reception of that care, and drug use and profiles. The SF-36 will be used to measure the general health component and quality of life of our sample (4). This will be a pragmatic study that will allow us the opportunity to develop further investigations leading to a larger scale and more robust clinical trial. In addition, this study will provide information on the challenges and opportunities involved in conducting clinical research concerning M/MT in a military setting and may lead to additional studies at a wider number of bases throughout the US.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty
* Aged 18-35
* New episode of low back pain (LBP) or a reoccurence of a past episode of low back pain

Exclusion Criteria:

* LBP from other somatic tissues as determined by history, examination, and course (i.e. pain referred from visceral conditions)
* Radicular pain worse than back pain
* Co-morbid pathology or poor health conditions that may directly impact spinal pain. Patients who have case histories and physical examination findings indicating other than average health will be excluded from the study
* Bone and joint pathology contraindicating patient for M/MT. Patients with spinal fracture, tumors, infections, inflammatory arthropathies and significant osteoporosis will be referred for appropriate care and will be excluded from the study
* Other contraindications for M/MT of the lumbar spine and pelvis (i.e. bleeding disorders or anticoagulant therapy)
* Pregnancy (all potential female participants will undergo pregnancy testing)
* Use of manipulative care for any reason within the past month
* Unable to follow course of care for four weeks
* Unable to give informed consent for any reason
* Unable to confirm that they will not be deployed during the course of the study: "Will you be deployed, receiving orders for a distant temporary active duty assignment, attending training at a distant sight, or otherwise absent from Ft. Bliss over the next 6 weeks?"

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Decreased pain | Baseline, 2 weeks, 4 weeks

SECONDARY OUTCOMES:
Increased function | Baseline, 2 weeks, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: CPT Keith P Myers, MD, Principal Investigator — William Beaumont Army Medical Center
Locations (1):
- Center for Integrative Medicine (CIM) at William Beaumont Army Medical Center; Soldier Family Medical Clinic (SFMC) at Ft. Bliss, TX, El Paso, Texas, United States

REFERENCES:
- [Derived] Goertz CM, Long CR, Hondras MA, Petri R, Delgado R, Lawrence DJ, Owens EF, Meeker WC. Adding chiropractic manipulative therapy to standard medical care for patients with acute low back pain: results of a pragmatic randomized comparative effectiveness study. Spine (Phila Pa 1976). 2013 Apr 15;38(8):627-34. doi: 10.1097/BRS.0b013e31827733e7. PMID 23060056